CLINICAL TRIAL: NCT06563674
Title: Nurse-led Acceptance-based Healthy Lifestyles Program for Community-dwelling Patients With Pneumoconiosis: A Waitlist Pilot Randomized Controlled Trial
Brief Title: Acceptance-based Healthy Lifestyles Program for Patients With Pneumoconiosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Lon Tam, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: temp
Record Dates: First submitted 2024-08-13; First posted 2024-08-21 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-08

CONDITIONS: Pneumoconiosis; Healthy Lifestyle
Keywords: Pneumoconiosis; Healthy Lifestyle; Acceptance-based
MeSH Terms: conditions — Pneumoconiosis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A 2-arm waitlist pilot randomized controlled trial will be adopted. After baseline data collection, participants in the intervention group will receive the health program for 6 weeks. On the other hand, participants in the waitlist-control group will receive the same health program week 8 and week 14.
Who Masked: Outcomes Assessor
Masking Description: The baseline data will be collected by research assistant (RA)1 before randomization, while the follow-ups data will be collected by RA2. The participant's group allocation is masked to the outcome assessors. But the participants know their group allocation after randomization because of the nature of the intervention. Different dates will be planned for different groups for all follow-ups respectively to avoid contamination of the subjects and blinding to the outcome assessors as far as possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Participants will receive the acceptance-based healthy lifestyles program between week 8-14.
  Interventions: Other: Acceptance-based healthy lifestyles program (control group)
- Intervention (Experimental): Participants will receive the acceptance-based healthy lifestyles program between week 1-6.
  Interventions: Other: Acceptance-based healthy lifestyles program (intervention group)

INTERVENTIONS:
Other: Acceptance-based healthy lifestyles program (intervention group) — The acceptance-based healthy lifestyles program consists of 4 biweekly 60-min face-to-face interactive workshops to cover the knowledge of pneumoconiosis, exercise to maintain lung function, health diet, and home safety.
  Arms: Intervention
Other: Acceptance-based healthy lifestyles program (control group) — The acceptance-based healthy lifestyles program consists of 4 biweekly 60-min face-to-face interactive workshops to cover the knowledge of pneumoconiosis, exercise to maintain lung function, health diet, and home safety.
  Arms: Control

SUMMARY:
Symptoms, such as cough and shortness of breath, are common among patients with pneumoconiosis. Depression and anxiety can be elicited by the symptoms, while avoidance of daily activities is believed to reduce trigger of symptoms. The lung function is then declined and the risk of having stroke and heart failure is increased. The objectives of this 2-arm waitlist pilot randomized controlled trial are to test the effects and feasibility of an acceptance-based educational program among patients with pneumoconiosis. 80 participants will be recruited from community centers and randomly assigned to intervention group or waitlist-control group in a ratio of 1:1. The 6-week group-based educational program will be provided to the intervention group first, then the waitlist-control group. The program consists of 4 sessions integrated with acceptance components and care of pneumoconiosis. Their psychological health, healthy lifestyles, and cardiometabolic profiles will be assessed at baseline, week 6, and week 14. Data will be analyzed using a statistical package. The feasibility of the program will be evaluated by interview. The findings of this study can inform the integration of acceptance-based intervention into pneumoconiosis management in Hong Kong, and future study on chronic progressive lung diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese who is able read and speak Chinese.
2. Adults aged 18 or over.
3. Taking compensation for pneumoconiosis.

Exclusion Criteria:

1. Those who have mental, visual, hearing, or cognitive impairments with regular medical follow-ups and treatment.
2. Those who are unable to give written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Psychological flexibility | Baseline, week 6, and week 14
  Measured by Acceptance and Action Questionnaire-II Chinese version. It is a 7-point Likert scale with 7 items. The score ranges from 7 to 49 and a higher total score indicates less flexibility.

SECONDARY OUTCOMES:
Exercise-related outcome | Baseline, week 6, and week 14
  Measured by Self-Efficacy for Exercise scale Chinese version The Chinese scale has 9 items, 11-point Likert scale. A higher total score indicates people have more self-efficacy to do exercise, range from 0 to 90.
Practice of healthy diet | Baseline, week 6, and week 14
  Measured by the diet subscale of the Chinese version of Health Promoting Lifestyle Profile II The subscale consists of 8 items to assess the practice of healthy diet. It is a 4-point Likert scale that a higher score indicates the more practice of healthy diet (range 8 to 32).
Blood pressure | Baseline, week 6, and week 14
  Measured by validated and reliable upper-arm automated system after resting for 20 min
Waist circumference | Baseline, week 6, and week 14
  Measured in nearest 0.1 centimeter
Body weight | Baseline, week 6, and week 14
  Measured by a calibrated digital body monitor with participants wearing similar light clothing without shoes and socks
Glycated hemoglobin (HbA1c) | Baseline and week 14
  blood test

CONTACTS AND LOCATIONS:
Locations (1):
- PMAA, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Available upon request and approval from the funding body.